CLINICAL TRIAL: NCT01340352
Title: Is It Possible to Predict Pre Term Labor by Measuring Cervical Length in the Non-pregnant Uterus?
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Etty Spiegel, Director of Ultrasound Unit, HaEmek Medical Center, Israel
Other Study IDs: 0137-10-EMC
Record Dates: First submitted 2011-04-20; First posted 2011-04-22 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- study group: previous preterm labor
- control group:previous term delivery

SUMMARY:
Working hypothesis and aims:

To investigate the association between cervical length in non-pregnant women, and the risk of premature birth.

The participants will be recruited from the HaEmek Medical Center delivery room registration. Women delivered between 24-37 pregnancy weeks will be allocated to the study group. The investigators will invite them 3 month or more after delivery to ultrasound examination of the cervical length. The participants in the control group will be the women whom term delivery follows by chronological manner to those in study group. Data of the cervucal length will be collected at the time of the examination.

DETAILED DESCRIPTION:
Women will be invited to undergo an examination in Ultrasound Unit of Department of Obstetrics and Gynecology, HaEmek Medical Center.

Ultrasound examination will be performed using the Voluson E8 device, General Electric.

The cervical length,between the external and internal orifice will be measured using conventional technologies available including: Doppler, three dimensional and two dimensional ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Nonpregnant women aged 18-40 years.
* Singelton last pregnancy.
* Last birth, spontaneous premature (24-37 week)
* Last birth at least 3 months ago.

Exclusion Criteria:

* Presence of uterine malformations.
* Sonographic pathologic findings.
* Technical failure (failed appropiate sonographic visualisation)
* Presence of fetal malformations ( in preterm delivery )
* Presence of comorbidities including diabetes, hypertension, collagen disease, thrombophilia
* Presence of risk factors for premature delivery (amniotic fluid infection,

  * cervical surgical treatments - conization, polyhydramnios, etc.).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: HaEmek Medical Center delivery room.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2011-05; Primary Completion 2012-05 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
length of the cervix in mm. | up to 20 month
  External orifice location is well-defined anatomically and easy for identification .Internal orifice location will be determined by the level of the uterine arteries at both sides of the cervix.

CONTACTS AND LOCATIONS:
Overall Officials: Etty Daniel-Spiegel, MD, Principal Investigator — haemek medical center
Locations (1):
- Dep. OB/GYN, Emek Medical Center, Afula, Israel